CLINICAL TRIAL: NCT00235235
Title: Predicting Response and Toxicity in Patients Receiving Chemotherapy for Breast Cancer: A Multicenter Genomic, Proteomic and Pharmacogenomic Correlative Study: Hoosier Oncology Group COE-01
Brief Title: A Correlative Study for Predicting Response and Toxicity in Patients Receiving Chemotherapy for Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Funding terminated
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Indiana University School of Medicine (Other); Walther Cancer Institute (Other)
Responsible Party: Principal Investigator, Kathy Miller, MD, Professor, IU School of Medicine, Hoosier Cancer Research Network
Other Study IDs: HOG COE-01; Department of Defense BC030400 (Registry Identifier: ClinicalTrials.Gov)
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy; Urine Specimen Collection; Doxorubicin; Cyclophosphamide; Capecitabine; Vinorelbine; Gemcitabine

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — core biopsy, serum, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- A: Doxorubicin 60 mg/m2 + Cyclophosphamide 600 mg/m2 day 2 of every 21-day cycle
  Interventions: Procedure: Biopsy; Procedure: Serum Collection; Procedure: Urine Collection; Drug: Doxorubicin; Drug: Cyclophosphamide
- B: Capecitabine 1000mg/m2 bid days 1-14 of every 21-day cycle
  Interventions: Procedure: Biopsy; Procedure: Serum Collection; Procedure: Urine Collection; Drug: Capecitabine
- C: Vinorelbine 25 mg/m2 days 1, 8, 15 of every 28-day cycle
  Interventions: Procedure: Biopsy; Procedure: Serum Collection; Procedure: Urine Collection; Drug: Vinorelbine
- D: Gemcitabine 1000mg/m2 days 1, 8, 15 of every 28-day cycle
  Interventions: Procedure: Biopsy; Procedure: Serum Collection; Procedure: Urine Collection; Drug: Gemcitabine

INTERVENTIONS:
Procedure: Biopsy — core biopsy
Procedure: Serum Collection — serum collection
Procedure: Urine Collection — urine collection
Drug: Doxorubicin — Doxorubicin 60 mg/m2 day 1 of every 21-day cycle
  Groups: A
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m2 day 1 of every 21-day cycle
  Groups: A
Drug: Capecitabine — Capecitabine 1000 mg/m2 bid days 1-14 of every 21-day cycle
  Groups: B
Drug: Vinorelbine — Vinorelbine 25mg/m2 days 1, 8, 15 of every 28-day cycle
  Groups: C
Drug: Gemcitabine — Gemcitabine 1000mg/m2 days 1, 8, 15 of every 28-day cycle
  Groups: D

SUMMARY:
The proposed trial provides a unique opportunity in that it combines genomic, proteomic, and pharmacogenomic assessments in patients receiving the most commonly used chemotherapies for advanced breast cancer. To date no other trial has analyzed gene and protein expression at the same time points in the same patient, combined with clinical outcome. Similar to previous attempts to predict response based on expression of a single gene or protein, the researchers expect that neither genomic or proteomic profiling alone will be sufficient to optimize therapy. Rather, the researchers expect an iterative process that combines information gleaned from both platforms, modified to avoid toxicity based on pharmacogenomics.

DETAILED DESCRIPTION:
OUTLINE: This is a 4 arm, multi-center study.

Sample Collection:

* Core Biopsy
* Serum
* Urine

Treatment Regimens (Investigator/Patient Discretion):

* Arm A: Doxorubicin 60 mg/m2 + Cyclophosphamide 600 mg/m2 day 1 of every 21-day cycle
* Arm B: Capecitabine 1000 mg/m2 BID days 1-14 of every 21-day cycle
* Arm C: Vinorelbine 25 mg/m2 days 1, 8, 15 of every 28-day cycle
* Arm D: Gemcitabine 1000 mg/m2 days 1, 8, 15 of every 28-day cycle

Performance status & Organ Function:

Performance status and organ function appropriate for chemotherapy in the opinion of the treating investigator according to Good Clinical Practice (GCP).

Life Expectancy: Not specified

Hematopoietic: Not specified

Hepatic: Not specified

Renal: Not specified

Cardiovascular: Not specified

Pulmonary: Not specified

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast with locally advanced or metastatic disease.
* Disease amenable to pre-treatment core or incisional biopsy with adequate tissue for histology and genomic/proteomic analysis.
* Measurable disease as assessed within 21 days prior to being registered for protocol therapy by RECIST.
* Planned chemotherapy with one of the following regimens:

  1. Doxorubicin 60 mg/m2 + Cyclophosphamide 600 mg/m2 day 1 of every 21-day cycle
  2. Capecitabine 1000 mg/m2 BID days 1-14 of every 21-day cycle
  3. Vinorelbine 25 mg/m2 days 1, 8, 15 of every 28-day cycle
  4. Gemcitabine 1000 mg/m2 days 1, 8, 15 of every 28-day cycle

Exclusion Criteria:

* No serious uncontrolled medical or surgical condition that the investigator feels might compromise study participation.
* Negative pregnancy test obtained within 7 days prior to being registered for protocol therapy for women of child bearing potential.
* Unwillingness to use adequate contraception (or practicing complete abstinence). Subjects should be advised that adequate contraception (or complete abstinence) must be continued while on treatment and for a period of 3 months after the final dose of chemotherapy.
* No breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study limited to patients with breast cancer.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To correlate tumor gene expression (genomic profile) with response to commonly used chemotherapies in patients with advanced breast cancer | 36 months

SECONDARY OUTCOMES:
To correlate serum and tumor proteomic profiles with response to commonly used chemotherapies. | 36 months
To compare serum and tissue proteomic analyses. | 36 months
To compare genomic and proteomic profiles. | 36 months
To correlate toxicity and/or response with drug-specific pharmacogenomic parameters. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, M.D., Study Chair — Hoosier Oncology Group, LLC; George Sledge, M.D., Principal Investigator — Hoosier Oncology Group, LLC
Locations (11):
- United States (10):
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Mary Lou Mayer, M.D., Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Baylor College of Medicine - Methodist Breast Center, Houston, Texas
- Instituto de Enfermedades Neoplasticas (INEN), Lima, Peru

REFERENCES:
- See also: Hoosier Oncology Group Home Page — http://www.hoosieroncologygroup.org